CLINICAL TRIAL: NCT01625299
Title: PILOT STUDY: The Physiological Basis for Dietary Protein Intolerance in Children With Autism
Brief Title: Pilot Study of Diet and Behavior in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Fernando Navarro, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSC-MS-07-0223
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Autism
Keywords: intestinal permeability; diet; gluten; dairy
MeSH Terms: conditions — Autistic Disorder | interventions — Glutens; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gluten and Milk group (Experimental): Subject on a gluten and dairy free diet will receive supplement of gluten and dry milk daily
  Interventions: Dietary Supplement: Gluten and dry milk
- Rice flour (Placebo Comparator): Subjects will be on a gluten and dairy free diet and receive daily supplement of rice flour (placebo)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Gluten and dry milk — 0.5 g/kg/day of gluten 0.5 g/kg/day of dry milk
  Other Names: Gluten and dairy group
  Arms: Gluten and Milk group
Dietary Supplement: Placebo — Rice flour 1.0 g/kg/day
  Other Names: Control group
  Arms: Rice flour

SUMMARY:
We hypothesize that in children with autism dietary antigens can change the intestine, making it "leaky" and then affecting the brain changing their behavior.

DETAILED DESCRIPTION:
Subjects in 2 different diets (gluten/dairy and placebo) will be monitored for changes in intestinal permeability (urine lactulose mannitol ratio) and behavior (psychometric testing).

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 3 and 12 years,
* DSM-IV (APA, 2000) diagnosis of Autistic Disorder (DSM-IV 299.90),
* willingness to follow and maintain a gluten-free-dairy-free-diet for 4 weeks.

Exclusion Criteria:

* food allergies,
* celiac disease,
* inflammatory bowel disease,
* infectious gastrointestinal,
* seizure disorder,
* neurological problems with behavioral changes,
* unwillingness to undertake the dietary challenge with milk and gluten or to maintain a gluten-free-dairy-free-diet during the study were excluded

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Intestinal Permeability | baseline, 2 weeks and 4 weeks
  Changes in intestinal permeability and behavior with changes in diet

SECONDARY OUTCOMES:
Psychometric testing | baseline, 2 weeks and 4 weeks
  Behavioral variables: hyperactivity, innatention, irritability
Gastrointestinal symptoms | baseline, week 2, week 4
  Changes in gastrointestinal symptoms with different diets

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Navarro, M.D>, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center At Houston, Houston, Texas, United States